CLINICAL TRIAL: NCT03337048
Title: Exploratory Study Investigating Urodynamic Parameters During Catheterisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP277
Record Dates: First submitted 2017-11-07; First posted 2017-11-08 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injuries; Enlarged Prostate With Lower Urinary Tract Symptoms
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement of endpoints (Experimental): In healthy volunteers the endpoint are measured while spontaneous voiding of the bladder and while emptying the bladder using a standard intermittent catheter.
  In subjects with spinal cord injury or enlarged prostata the endpoint are measured while emptying the bladder using a standard intermittent catheter.
  Interventions: Device: SpeediCath

INTERVENTIONS:
Device: SpeediCath — SpeediCath is a standard intermittent catheter that is on the market.

SUMMARY:
The objective of the study is to explore and understand how urodynamic parameters are affected when emptying the bladder with an intermittent catheter.

DETAILED DESCRIPTION:
The investigation is an explorative open single arm investigation including 30 male subjects. 10 healthy volunteers, 10 patients with SCI and 10 patients with BPH.

The healthy volunteers included into the study will have an information visit and three study visits - an inclusion visit (visit 0), a visit 1 measuring endpoints while spontaneous voiding of the bladder (0-7 days after visit 0) followed by a visit 2 measuring endpoints while emptying the bladder using a standard IC (4-15 days after visit 1). (Visit 0 and visit 1 can be the same day).

The subjects with SCI and enlarged prostate will have an information visit and two study visits. - an inclusion visit (visit 0) where a urine culture is analysed and prophylactic antibiotic is prescribed per the result of the analysis. (Most IC users have bacteria in the urine and to decrease the risk of acquiring a urinary tract infection from the urodynamic examination, urine cultures are performed and prophylactic antibiotics will be prescribed per the result). The second visit (visit 1) is conducted while the patient is on antibiotic treatment measuring all endpoints while emptying the bladder with a standard IC (4-15 days after visit 0 while subject is on prophylaxis antibiotics).

The investigation is conducted at one site and is an explorative study, estimated to last eight (8) months.

Due to the explorative nature of the investigation, no primary endpoint is defined but explorative endpoints are divided into three categories dependent on their relation to bladder, urethra or urine.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent
2. Be at least 18 years of age and have full legal capacity
3. Be male
4. For healthy volunteers: Willing to comply with not using analgesics up to 24 hours prior to study visit
5. For healthy volunteers: Negative urine multistix (leukocytes and nitrite), or if positive, subsequent negative for bacterial growth in urine culture
6. For SCI and BPH patients: Use intermittent catheter daily and have used intermittent catheters for at least 2 months

Exclusion Criteria:

1. Symptoms of urinary tract infections (frequent urination, stinging and pain at urination)
2. Participate in other clinical investigations related to urinary tract system during this investigation (Inclusion → termination)
3. For healthy volunteers: Abnormalities, diseases or surgical procedures performed in the lower urinary tract

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male subjects are included as the intermittent catheter used in the investigation is a male catheter
Enrollment: 30 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazarena Mazarro, Study Director — Vice president Medical Affairs
Locations (1):
- Department of Urology, Rigshospitalet, Copenhagen, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: 10 healthy volunteers
- Spinal Cord Injury (SCI): 10 spinal cord injured patients
- Benign Prostate Hyperplasia: 10 benign prostate hyperplasia patients
Period: Overall Study
Arm/Group | Healthy Volunteers | Spinal Cord Injury (SCI) | Benign Prostate Hyperplasia
Started | 10 | 10 | 10
Completed | 8 | 10 | 10
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Urodynamic Parameters During Catheterisation: Exploratory measurements of Urodynamic parameters
Arm/Group | Urodynamic Parameters During Catheterisation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 30

OUTCOME MEASURES:

1. Primary Outcome: Discomfort During Catheter Insertion on a Visual Analogue Scale
Description: On a scale ranging from 0 "no discomfort" to 10 "worst possible discomfort" caused by the catheter, set a vertical line indicating how you experienced the insertion of the catheter. Higher scores mean a worse outcome.
Time Frame: Filled out after 5 minutes per catheterisation.
Population: 8 healthy volunteers, 10 subjects with spinal cord injury and 10 subjects with enlarged prostate
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Measurement of Endpoints: In healthy volunteers the endpoint are measured while spontaneous voiding of the bladder and while emptying the bladder using a standard intermittent catheter (SpeediCath).
  In subjects with spinal cord injury or enlarged prostata the endpoint are measured while emptying the bladder using a standard intermittent catheter.
  SpeediCath: SpeediCath is a standard intermittent catheter that is on the market.
Arm/Group | Measurement of Endpoints
Number analyzed (Participants) | 28
score on a scale
  healthy volunteers: number analyzed (Participants) | 8
  healthy volunteers | 1.2 [0.1 to 3.9]
  Spinal Cord Injury: number analyzed (Participants) | 10
  Spinal Cord Injury | 1.0 [0.0 to 6.1]
  Benign prostatic hyperplasia: number analyzed (Participants) | 10
  Benign prostatic hyperplasia | 1.1 [0.0 to 2.6]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 15 days.
Description: An adverse event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other parties, whether related to the medical device(s), or the procedures involved or not. This could include events such as headache or dizziness.
Arm/Group | Measurement of Endpoints
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT03337048/Prot_SAP_000.pdf